CLINICAL TRIAL: NCT00931073
Title: A Phase I, Open-Label, Three-Period, Fixed-Sequence Study To Estimate The Steady-State Effect Of Ketoconazole And Omeprazole On The Single-Dose Pharmacokinetics Of Dimebon [PF-01913539] In Healthy CYP2D6 EM And PM Subjects
Brief Title: A Phase I Study To Estimate The Effect Of Ketoconazole And Omeprazole On The Pharmacokinetics Of Dimebon In Healthy Subjects Who Are Normal Or Poor CYP2D6 Metabolizers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: B1451017
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Alzheimer's Disease; Huntington's Disease
Keywords: Drug Interactions; pharmacokinetics; CYP2D6; CYP2C19; ketoconazole; omeprazole
MeSH Terms: conditions — Alzheimer Disease; Huntington Disease | interventions — latrepirdine; Ketoconazole; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Period 1 (Experimental)
  Interventions: Drug: Dimebon alone
- Period 2 (Experimental)
  Interventions: Drug: Dimebon + Ketoconazole
- Period 3 (Experimental)
  Interventions: Drug: Dimebon + Omeprazole

INTERVENTIONS:
Drug: Dimebon alone — Pharmacokinetics of a single oral dose of 10 mg Dimebon (tablet) will be assessed in subjects with a CYP2D6 extensive and poor metabolizer status based on genotyping as screening
  Arms: Period 1
Drug: Dimebon + Ketoconazole — Pharmacokinetics of a single oral dose of 10 mg Dimebon (tablet) will be assessed on Day 4 during the daily administration of ketoconazole (400 mg, Day 1-11) in subjects with a CYP2D6 extensive and poor metabolizer status based on genotyping as screening
  Arms: Period 2
Drug: Dimebon + Omeprazole — Pharmacokinetics of a single oral dose of 10 mg Dimebon (tablet) will be assessed on Day 5 during the daily administration of omeprazole(40 mg, Day 1-12) in subjects with a CYP2D6 extensive and poor metabolizer status based on genotyping as screening
  Arms: Period 3

SUMMARY:
This study will evaluate the potential for a drug-drug interaction of Dimebon with ketoconazole and omeprazole, potent inhibitors of the drug metabolizing enzymes CYP3A4 and CYP2C19, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Subjects must have either a CYP2D6 EM (n=12) or PM (n=12) status based on genotyping at screening.
* Subjects must have a CYP2C19 EM status based on status at screening.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Subjects with any history of a previous seizure or convulsion or significant head trauma.
* Subjects specifically allergic to imidazole antifungal agents.
* Subjects specifically allergic to omeprazole or other proton pump inhibitors.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Subjects with hypersensitivity reactions to Dimebon or other antihistamines.
* Consumption of grapefruit or grapefruit containing products within 7 days prior to the first dose of study medication.
* Subjects currently taking omeprazole, other proton pump inhibitors, antacids, H2-blockers or CYP2C19 inhibitors.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of nonhormonal contraception as outlined in this protocol from at least 14 days prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Dimebon alone: Dimebon PK in CYP2D6 EMs and PMs (Cmax, Tmax, AUCinf (as data permit), AUClast, and t1/2 (as data permit), CL/F (as data permit) and V/F (as data permit)) | Period 1 Day 1
Dimebon + keto: Dimebon PK in CYP2D6 EMs and PMs (Cmax, Tmax, AUCinf (as data permit), AUClast, and t1/2 (as data permit), CL/F (as data permit) and V/F (as data permit)) | Period 2 Day 4
Dimebon + omeprazole: Dimebon PK in CYP2D6 EMs and PMs (Cmax, Tmax, AUCinf (as data permit), AUClast, and t1/2 (as data permit), CL/F (as data permit) and V/F (as data permit)) | Period 3 Day 5

SECONDARY OUTCOMES:
Dimebon alone: Safety and tolerability (AE's, ECG, vital signs, safety labs) | Period 1 Day 1-7
Dimebon + keto: Safety and tolerability (AE's, ECG, vital signs, safety labs) | Period 2 Day 1-12
Dimebon + omeprazole: Safety and tolerability (AE's, ECG, vital signs, safety labs) | Period 3 Day 1-13

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Kalamazoo, Michigan, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451017&StudyName=A%20Phase%20I%20Study%20To%20Estimate%20The%20Effect%20Of%20Ketoconazole%20And%20Omeprazole%20On%20The%20Pharmacokinetics%20Of%20Dimebon%20In%20Healthy%20Subjects%20Who%20Are